CLINICAL TRIAL: NCT05113420
Title: The Efficacy and Safety of Different Phlebotonic Drugs in Children With Venous Malformations: a Prospective Cohort Study
Brief Title: The Efficacy and Safety of Different Phlebotonic Drugs in Children With Venous Malformations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Vascular Pathology, Moscow (Other)
Responsible Party: Sponsor
Other Study IDs: VAC_VM
Record Dates: First submitted 2021-10-09; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Drug Effect; Children, Only; Vascular Malformations; Surgery
MeSH Terms: conditions — Vascular Malformations | interventions — S 5682; troxevasin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Per os+topical solution(1)
  Interventions: Drug: Detralex
- Per os+topical solution(2)
  Interventions: Drug: Detralex; Drug: Troxevasin
- Per os only
  Interventions: Drug: Detralex
- Topical solution only
  Interventions: Drug: Detralex; Drug: Troxevasin

INTERVENTIONS:
Drug: Detralex — Diosmin+ Hesperidin
Drug: Troxevasin — Troxerutin
  Groups: Per os+topical solution(2); Topical solution only

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of different phlebotonic drugs in children and to assess patient satisfaction after treatment.

ELIGIBILITY:
Inclusion Criteria: venous malformation

* venous malformation

Exclusion Criteria:

* allergy

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-11-17 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
Coagulation testing | 1 month
  Coagulation testing

OTHER OUTCOMES:
Satisfaction after treatment | 1 month
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Listovskaia, MD, Study Chair — Vascular Anomalies Center (VAC) "Hemangioma" LLC.; Dmitriy Romanov, MD, Study Chair — Vascular Anomalies Center (VAC) "Hemangioma" LLC.
Locations (1):
- The Vascular Anomalies Center (VAC) "Hemangioma" LLC, Moscow, Russia